CLINICAL TRIAL: NCT04088747
Title: Logistic Regression and Elastic Net Regularization for the Diagnosis of Fibromyalgia: A Quantitative Approach Using B-Mode Ultrasound
Brief Title: Logistic Regression and Elastic Net Regularization for the Diagnosis of Fibromyalgia
Acronym: LEDF
Status: Completed | Type: Observational
Sponsor: Toronto Rehabilitation Institute (Other)
Responsible Party: Principal Investigator, Dinesh Kumbhare, Affiliate Scientist, Toronto Rehabilitation Institute
Other Study IDs: FibromyalgiaDiagnosis
Record Dates: First submitted 2019-09-11; First posted 2019-09-13 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Ultrasound; Regularization; Logistic Regression; Imaging
MeSH Terms: conditions — Fibromyalgia | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fibromyalgia: Patients who display symptoms and have a history of Fibromyalgia, between 20-65 years of age.
  Interventions: Diagnostic Test: Ultrasound Imaging
- Healthy Controls: Age-matched, healthy controls, between 20-65 years of age who present no signs of chronic pain.
  Interventions: Diagnostic Test: Ultrasound Imaging

INTERVENTIONS:
Diagnostic Test: Ultrasound Imaging — B-mode ultrasound pictures of the upper Trapezius were collected from both left and right sides.

SUMMARY:
This study will utilize ultrasound image texture variables to construct an elastic net regularized, logistic regression model to differentiate between healthy and Fibromyalgia patients. The collected ultrasound data will be from participants who are healthy, and from participants who have Fibromyalgia. The predicted performance accuracy of the diagnostic model will be validated and this will confirm or deny the hypothesis that differentiation between the two cohorts is possible.

DETAILED DESCRIPTION:
Fibromyalgia (FM) diagnosis remains a challenge for clinicians due to a lack of objective diagnostic tools. One proposed solution is the use of quantitative ultrasound (US) techniques, such as image texture analysis, which has demonstrated discriminatory capabilities with other chronic pain conditions. The investigators propose the use of US image texture variables to construct an elastic net regularized, logistic regression model, for differentiating between the trapezius muscle in the healthy and FM patients. 162 Ultrasound videos of the right and left trapezius muscle were acquired from healthy participants and participants with FM. The videos will then be put through a mutli-step processing pipe including converting them into skeletal muscle regions of interest (ROI). The ROI's will be then filtered by an algorithm utilizing the complex wavelet structural similarity index (CW-SSIM), which removes ROI's that are too similar to one another. Eighty-eight texture variables will be extracted from the ROI's, which will be used in nested cross-validation to construct a logistic regression model with and without elastic net regularization. The generalized performance accuracy of both models will be estimated and confirmed with a final validation on a holdout test set. Depending on the predicted, generalized performance accuracy it will be validated or not by the final, holdout test set (confirming the model construction is accurate). These models should then confirm or deny the hypothesis that a regularized logistic regression model built on ultrasound texture features can accurately differentiate between healthy trapezius muscle and that of patients with FM.

ELIGIBILITY:
Inclusion Criteria:

* gender independent; chronic widespread pain, fitting the 2016 FM criteria, absence of myofascial pain syndrome trigger points and between the ages of 20 and 65 years (44.3 ± 13.9 years).
* Healthy asymptomatic volunteers who were age matched (n = 17) with no physical complaints or abnormality on physical examination also participated.

Exclusion Criteria:

* Participants were excluded if they demonstrated clinical evidence of another cause for widespread pain, such as polymyositis, dermatomyositis, endocrine disorders, etc. None of the participants had performed any physical exercise during the two to three days prior to entry into the study.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Fibromyalgia and healthy age-matched controls.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2019-09-06 (Actual)

PRIMARY OUTCOMES:
Ultrasound Image Texture Variables | 1 hour
  91 statistical image texture variables are extracted from the B mode ultrasound images from both cohorts in order to construct a diagnostic model. The texture variables will be extracted using MATLAB.
Fibromyalgia Diagnostic Criteria | 10 minutes
  This evaluates symptoms related to Fibromyalgia and determines a score to assess the severity. This score is comprised of the Widespread Pain Index(WPI), which quantifies the regions of pain, and the Symptom Severity Scale(SSS), which measures qualitative aspects of pain such as fatigue and cognitive symptoms. The WPI scale ranges from 0-19 (0- no areas of body pain, 19- all body regions have pain), whereas the SSS ranges from 0-12 (0-no qualitative aspects of pain, 12-many qualitative aspects of pain). This criteria was evaluated on each patient to determine which cohort they belong to. According to the Fibromyalgia Diagnostic Criteria, one is diagnosed with Fibromyalgia if they have a WPI score of 7 or higher, and a SSS score of 5 or higher. Fibromyalgia is also diagnosed with a score of 3-6 on the WPI score, and a score of 9 or higher on the SSS score.
Central Sensitization Inventory | 10 minutes
  This is a self reported outcome measure designed to identify patients that experience central sensitization. It involves 25 questions which include symptomatic experiences. The subject must answer on a scale of 0(never) to 5(always) corresponding to how often they experience these. The maximum score is 100 and a score of more than 40 indicates the presence of Central Sensitization. This criteria was evaluated on each patient to determine which cohort they belong to.

CONTACTS AND LOCATIONS:
Overall Officials: Dinesh Kumbhare, MD,PhD, Principal Investigator — Toronto Rehabilitation Institute
Locations (1):
- Toronto Rehabilitation Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wolfe F, Ross K, Anderson J, Russell IJ, Hebert L. The prevalence and characteristics of fibromyalgia in the general population. Arthritis Rheum. 1995 Jan;38(1):19-28. doi: 10.1002/art.1780380104. PMID 7818567
- [Background] Gittins R, Howard M, Ghodke A, Ives TJ, Chelminski P. The Accuracy of a Fibromyalgia Diagnosis in General Practice. Pain Med. 2018 Mar 1;19(3):491-498. doi: 10.1093/pm/pnx155. PMID 29016895
- [Background] Schaefer C, Mann R, Masters ET, Cappelleri JC, Daniel SR, Zlateva G, McElroy HJ, Chandran AB, Adams EH, Assaf AR, McNett M, Mease P, Silverman S, Staud R. The Comparative Burden of Chronic Widespread Pain and Fibromyalgia in the United States. Pain Pract. 2016 Jun;16(5):565-79. doi: 10.1111/papr.12302. Epub 2015 May 16. PMID 25980433
- [Background] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Hauser W, Katz RL, Mease PJ, Russell AS, Russell IJ, Walitt B. 2016 Revisions to the 2010/2011 fibromyalgia diagnostic criteria. Semin Arthritis Rheum. 2016 Dec;46(3):319-329. doi: 10.1016/j.semarthrit.2016.08.012. Epub 2016 Aug 30. PMID 27916278
- [Background] Ablin JN, Wolfe F. A Comparative Evaluation of the 2011 and 2016 Criteria for Fibromyalgia. J Rheumatol. 2017 Aug;44(8):1271-1276. doi: 10.3899/jrheum.170095. Epub 2017 Jun 1. PMID 28572464
- [Background] U.S. Department of Health and Human Services Food and Drug Administration/Centre for Drug Evaluation and Research. Guidance for Industry and FDA Staff Qualification Process for Drug Development Tools. Silver Spring, MD: Author; 2014
- [Background] Kravis MM, Munk PL, McCain GA, Vellet AD, Levin MF. MR imaging of muscle and tender points in fibromyalgia. J Magn Reson Imaging. 1993 Jul-Aug;3(4):669-70. doi: 10.1002/jmri.1880030418. PMID 8347962
- [Background] Meenagh G, Sakellariou G, Iagnocco A, Delle Sedie A, Riente L, Filippucci E, Di Geso L, Grassi W, Bombardieri S, Valesini G, Montecucco C. Ultrasound imaging for the rheumatologist XXXIX. Sonographic assessment of the hip in fibromyalgia patients. Clin Exp Rheumatol. 2012 May-Jun;30(3):319-21. Epub 2012 Jun 26. PMID 22734970
- [Background] Bendtsen L, Norregaard J, Jensen R, Olesen J. Evidence of qualitatively altered nociception in patients with fibromyalgia. Arthritis Rheum. 1997 Jan;40(1):98-102. doi: 10.1002/art.1780400114. PMID 9008605
- [Background] Kumbhare DA, Ahmed S, Behr MG, Noseworthy MD. Quantitative Ultrasound Using Texture Analysis of Myofascial Pain Syndrome in the Trapezius. Crit Rev Biomed Eng. 2018;46(1):1-31. doi: 10.1615/CritRevBiomedEng.2017024947. PMID 29717675
- [Background] MathWorks. Image Processing Toolbox., Release 2018a, The MathWorks Inc.,Natick, Massachusetts, United States
- [Background] Sampat MP, Wang Z, Gupta S, Bovik AC, Markey MK. Complex wavelet structural similarity: a new image similarity index. IEEE Trans Image Process. 2009 Nov;18(11):2385-401. doi: 10.1109/TIP.2009.2025923. Epub 2009 Jun 23. PMID 19556195
- [Background] Behr M, Noseworthy M, Kumbhare D. Feasibility of a Support Vector Machine Classifier for Myofascial Pain Syndrome: Diagnostic Case-Control Study. J Ultrasound Med. 2019 Aug;38(8):2119-2132. doi: 10.1002/jum.14909. Epub 2019 Jan 7. PMID 30614553
- [Background] Haralick, R. M., & Shanmugam, K. Textural features for image classification. IEEE Transactions on systems, man, and cybernetics. 1973;SMC-3(6):610-621.
- [Background] Galloway, M. M. Texture classification using gray level run length. Computer graphics and image processing. 1975;4(2):172-179.
- [Background] Zou, H., & Hastie, T. Regularization and variable selection via the elastic net. Journal of the royal statistical society: series B (statistical methodology) 2005;67(2):301-320.
- [Background] MathWorks. Statistics and Machine Learning Toolbox., Release 2018a, The MathWorks Inc.,Natick, Massachusetts, United States
- [Background] Jalalian A, Mashohor SB, Mahmud HR, Saripan MI, Ramli AR, Karasfi B. Computer-aided detection/diagnosis of breast cancer in mammography and ultrasound: a review. Clin Imaging. 2013 May-Jun;37(3):420-6. doi: 10.1016/j.clinimag.2012.09.024. Epub 2012 Nov 13. PMID 23153689
- [Background] Virmani, J., Kumar, V., Kalra, N., & Khandelwal, N. Prediction of liver cirrhosis based on multiresolution texture descriptors from B-mode ultrasound. International Journal of Convergence Computing 2013;1(1):19-37.
- [Background] Xian, G. M. An identification method of malignant and benign liver tumors from ultrasonography based on GLCM texture features and fuzzy SVM. Expert Systems with Applications 2010;37(10):6737-6741.
- [Background] Bishop, C. M. Pattern recognition and machine learning. New York, NY: Springer-Verlag: 2006. p. 205-207.
- [Background] Sarle, W. S. Stopped training and other remedies for overfitting. Computing science and statistics, 1996:352-360.

DOCUMENTS (1):
  • Study Protocol (2019-09-09): https://cdn.clinicaltrials.gov/large-docs/47/NCT04088747/Prot_001.pdf